CLINICAL TRIAL: NCT04803656
Title: Pulmonary Functions and Peripheral Muscle Strength and Their Relationship With Disease Duration and Prognosis in Patients With Different COPD Stages
Brief Title: Assessment of Pulmonary Functions and Peripheral Muscle Strength of COPD Patients in Different GOLD Stages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SAG-C-YLP-131217-0652
Record Dates: First submitted 2021-03-09; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Copd
Keywords: COPD; Pulmonary functions; Respiratory muscle strength; Peripheral muscle strength
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: COPD patients: Respiratory muscle strength, peripheral muscle strength in both upper and lower extremity were evaluated. Pulmonary function tests obtained during routine controls of patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assesment (Other): Demographic information of all subjects (age, gender, educational status, occupation, body weight, height, body mass index), clinical (diagnosis period) and medical status, personal history and family history, COPD stage, COPD Assessment Test (CAT) score, emergency and hospital admissions numbers in the last 3 months, exacerbation and hospitalization numbers in the last one year were recorded. Respiratory and peripheral muscle strengths are evaluated. Also pulmonary functions test results obtained.
  Interventions: Other: Assessment of COPD patients

INTERVENTIONS:
Other: Assessment of COPD patients — Assessments explained in the arm section were made as described in one session.

SUMMARY:
The purpose of this research was to examine the respiratory functions, respiratory muscle strength and peripheral muscle strength of patients with COPD in different groups and to evaluate their correlation with the duration and prognosis of the disease in COPD.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a common disease characterized by airway obstruction against harmful particles and gases in the airway and lungs, and is progressive, treatable and preventable.

The severity of the disease in COPD is determined according to the GOLD (Global Initiative for Chronic Obstructive Lung Disease) guidelines (2). While determining the severity of airway obstruction with the patient's spirometric values in COPD; Combined COPD assessment is made with symptomatic evaluation, number of exacerbations and hospitalizations. Airway restriction is numerically (GOLD 1-4), symptom evaluation and exacerbation risk combined with letter grouping (Group A-D).

There is a loss of respiratory and peripheral muscle strength in COPD patients. A mixture of various local and systemic causes was responsible for respiratory muscle dysfunction in COPD. Immobility, systemic inflammation, hypoxia of the tissue, oxidative stress and increased apoptosis of the skeletal muscle have been identified as possible pathogenic factors for loss of peripheral muscle strength in COPD patients.

it was aimed to evaluate the respiratory functions, respiratory muscle strength and peripheral muscle strength of patients with different COPD groups clinically and to evaluate their correlation with the duration and prognosis of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Being in COPD stable period and over the age of 40,
* The absence of abnormal laboratory findings,
* Not having a mental problem that prevents filling the questionnaires to be used in the study, - The absence of any other respiratory disease such as asthma,
* Giving the informed consent.

Exclusion Criteria:

* COPD exacerbation (hospitalization with acute exacerbation in the last 15 days),
* Presence of cognitive impairment,
* Pregnancy status,
* Ischemic heart disease,
* Kyphoscoliosis and advanced postural disorder,
* Orthopedic problems and amputation surgery,
* Emphysema, bullous lung disease,
* Presence of bronchiectasis,
* Previous thoracic surgery history,
* Presence of lung cancer,
* Advanced heart failure.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Respiratory Muscle Strength | 10 minutes after obtaining socio-demographic information (It was done between the 10th and 20th minutes of the assessment).
  It is a non-invasive test that indirectly demonstrates respiratory muscle strength with maximal inspiratory pressure (PImax) and maximal expiratory pressure (PEmax).Test were carried out according to American Thoracic Society (ATS) / European Respiratory Society (ERS) criteria.
Peripheral Muscle Strength Assessment-Upper extremity | 25 minutes after obtaining socio-demographic information. After the respiratory muscle strength evaluation, the patients were rested for 5 minutes (It was done between the 25th and 35th minutes of the assessment).
  Upper extremity: For grip strength test a manual hydraulic dynamometer was used according to the recommendations of the American Association of Hand Therapists (AETD). The patients were measured in sitting position, shoulder adduction at 90 °, elbow flexion, forearm in pronosupination, neutral and wrist joints in neutral position. Three consecutive measurements were obtained by giving 60-second rest breaks between measurements. The result obtained from the average of three measurements was recorded.
Peripheral Muscle Strength Assessment-Lower extremity | 40 minutes after obtaining socio-demographic information. After Upper extremity muscle strength evaluation patients were rested for five minutes (It was done between the 40th and 55th minutes of the assessment)
  M. Quadriceps femoris strength was evaluated for knee extension. M. Hamstring strength was evaluated for knee flexion. The test was applied with the "make test" technique that requires isometric contraction. Participant was asked to maintain maximum isometric contraction for 5 seconds, and the average of 3 consecutive maximum contraction measurements performed at 30-second intervals was recorded.
Pulmonary Function Test (PFT) results | 55 minutes after obtaining socio-demographic information.
  The PFT results of patients' performed during their routine controls taken into consideration. The percentages of the predicted values (percent) for forced expiratory volume in one second (FEV1), forced vital capacity (FVC), FEV1/FVC, mid-expiratory flow rate (MEF25-75) and peak expiratory flow (PEF) were used for statistical analysis.

SECONDARY OUTCOMES:
Duration of the disease | After the permission of patients, in the first 10 minutes of assessment while obtaining socio-demographic information of patients.
  Diagnosis year of the patient were recorded.
Exacerbation numbers in last one year | After the permission of patients, in the first 10 minutes of assessment while obtaining socio-demographic information of patients.
  Exacerbation numbers in last one year of the patients were recorded.
Hospitalization numbers in last one year | After the permission of patients, in the first 10 minutes of assessment while obtaining socio-demographic information of patients.
  Hospitalization numbers in last one year of the patients were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Begum Unlu, PT, MSc, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No